CLINICAL TRIAL: NCT06635642
Title: Auditory Research in Children Living With HIV Exposure-uninfected (ARCHIVE)
Acronym: ARCHIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: University of Kentucky (Other); University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Peter Torre, Professor, San Diego State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1 R01 DC022822-01
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dichotic Interaural Intensity Difference Training (Experimental)
  Interventions: Behavioral: Dichotic Interaural Intensity Difference (DIID) Training

INTERVENTIONS:
Behavioral: Dichotic Interaural Intensity Difference (DIID) Training — A total of five trials will be presented in a sequence and there will be 10 sequences per training session. Each of the 25 consonant-vowel-consonant words or digits 1 through 10 (excluding 7) will be presented to each ear during the session. The pairs will be randomized every time, and a word will never be paired with itself. After a sequence is completed, the difficulty of the task will be adjusted, in real time, based on performance on the prior task. If the child scored 4 or 5 of 5 correct in the poorer ear, then the IID will be decreased by 2 dB making the task more difficult. If the child scores 0, 1, or 2 of 5 correct, then the IID will be increased by 2 dB making the task easier. Last, if the child scores 3 of 5 correct, then the IID will remain unchanged for the next sequence.

SUMMARY:
To evaluate the association of in utero antiretroviral therapy (ART) exposure and hearing abilities of children who were perinatally HIV-exposed, but HIV-free, stratified by timing of maternal ART initiation.

DETAILED DESCRIPTION:
This is a non-randomized, cross-sectional study of 7-10-year-old children that will also include an observational (pre-post) clinical trial for those children who will require intervention. Children/parent pairs will be contacted during their 7-year-old visit as part of the Healthy Child Study (HCS). Collaborators include investigators from the HCS trial. They will assist in the recruitment and data sharing of children with perinatally exposed to HIV, but HIV-free (PHEF) and children HIV-unexposed and HIV-free (HUF) from the HCS. All personnel conducting the assessments will be blinded to the child's HIV exposure status. All peripheral measures of hearing (i.e., otoscopy, tympanometry, distortion product otoacoustic emissions [DPOAEs], and pure-tone audiometry) are routinely performed in clinic. Central auditory processing measures (i.e., dichotic digits testing [DDT] and speech recognition in noise) are not part of routine audiological evaluation but will not require any additional training since these measures are within the scope of work for pediatric clinical audiologists.

Audiological Evaluation: The hearing examination consists of questionnaire, otoscopy, tympanometry, pure-tone air-conduction and bone-conduction audiometry, speech recognition thresholds (SRTs), speech recognition in noise, DDT, and DPOAEs. Questionnaires, otoscopy, and tympanometry can be completed in clinic rooms but pure-tone audiometry, SRTs, DDT, speech recognition in noise, and DPOAEs will be completed in sound treated rooms. The hearing examination portion will take 60 minutes and children will be given breaks when needed. A detailed explanation of the procedures is outlined below.

Questionnaire: The detailed hearing-related health questionnaire will be administered to all participants. Questions will include: whether the child had a newborn hearing screening test, and if so, these data will be extracted from medical records to determine if they passed or failed; history of middle ear involvement; trauma to the ear(s) or head; family history of hearing loss and any other medical-related hearing history, mother/caregiver-perception of any hearing problems, noise exposure, and any previous hearing aid use. The demographic questions will include date of birth, sex, race, primary language spoken, educational level of the child, child's performance at school, caregiver's education level, occupational status, annual income, and family history of hearing loss.

Otoscopy and Tympanometry: In a designated clinic room within the Speech Therapy & Audiology Clinic at Tygerberg Hospital, an audiologist will perform an otoscopic evaluation on each ear of the child. Information about the presence of debris (e.g., cerumen) in the external ear canal, color and position of the eardrum, and presence/absence of a perforation will be noted. Tympanometry will then be performed by the audiologists. This provides information regarding the functioning of the tympanic membrane. The tympanogram will be a critical component to this proposal, because these measures will most likely identify otitis media in children and poor middle ear function will have a negative, but temporary effect on DPOAEs. If there is an active middle ear involvement based on otoscopy and tympanometry measures, testing will be discontinued, the child will be referred to the Ear, Nose and Throat (ENT) clinic within Tygerberg Hospital, and the child will be rescheduled for testing once the fluid/infection has been resolved and tympanometry is within normal limits.

Pure-tone Hearing Testing: An audiologist will perform all pure-tone audiometric testing using traditional assessment protocols. Pure-tone audiometry using supra-aural earphones will be completed. Testing will be conducted in a sound-treated booth on calibrated equipment. Air conduction (AC) thresholds will be obtained at octave frequencies from 0.25-8 kHz bilaterally. Masking will be used when appropriate. If AC thresholds are >15 decibels of hearing level (dB HL), a bone conduction (BC) transducer will be placed on the mastoid of the poorer ear, as determined by the air-conduction thresholds. BC thresholds will be determined at 0.5-4 kHz. If air bone gaps are noted, masking to obtain BC thresholds will be used at all frequencies with an air-bone gap ≥15 dB HL.

Distortion Product Otoacoustic Emissions: DPOAEs will be used to assess integrity of cochlear outer hair cell function. DPOAEs will be measured using two primary frequencies (f1 and f2, where f2 > f1) at f2/f1 = 1.22, f2 swept from 1 through 8 kHz, and a f1 level (L1) of 65 dB of sound pressure level (SPL) and a f2 level (L2) of 55 dB SPL. The child will be instructed to remain as quiet as possible and that they do not need to respond.

Speech Recognition Thresholds: SRT data will be obtained under earphones once pure-tone testing has been completed. The South African Spondaic wordlist will be presented in English and the lowest dB HL level that the child can repeat words 50% correctly will establish the SRT for each ear. Speech recognition in noise testing will then be completed. Presentation level of words will be determined as 50 dB above the SRT for each ear. For example, if the SRT for the right ear was 15 dB HL, then the fixed presentation level for that ear during speech recognition in noise would be 65 dB HL. This ensures a comfortable listening level well above the child's hearing thresholds. The background noise will be set 8 dB HL below the presentation level of the words. And in the example above, the background noise would be set to 57 dB HL. This is a more complex listening setting, but not too difficult for the children to be able to repeat the words that they hear.

Dichotic Digits Testing: DDT will be completed in order to evaluate binaural integration. Testing will be completed under earphones once the SRT has been established. The test will be presented at 50 dB above the SRT, consistent with speech recognition in noise, to ensure a comfortable listening level. The child will be instructed that they will hear two numbers in each ear simultaneously and to listen carefully in both ears and repeat all of the numbers they hear. The repeated order will not matter and guessing the numbers is acceptable. The child will be given practice items before scoring begins. The test will consist of 20 stimulus presentations, or 80 total digits (40 per ear). Numbers between 1-10 (with the exception of 7 due to not being monosyllabic) will be presented in a random order. Scoring for each ear will be calculated as percent correct for each ear.

Intervention: Children who meet the criterion for DDT deficit (>15% difference between the ears) will be scheduled for 12 Dichotic Interaural Intensity Difference (DIID) training sessions, 20-30 minutes each over a 4-6 week period. Training will take place in the afternoon at the FAMCRU satellite research unit in Khayelitsha, Michael Mapongwana Hospital, which is close to participants homes. Training will be administered using a custom iPad application routed through earphones within a quiet room at FAMCRU satellite research unit. Training will focus on the poorer ear as reflected on DDT scores. The training stimuli are a combination of English digits or consonant-vowel-consonant (CVC) words recorded by a male talker. The dichotic listening tasks focused on binaural integration only. Prior to starting the DIID training, the child's crossover point will be established. The crossover point is the interaural intensity difference (IID) during a dichotic task at which performance in the poorer ear exceeds the better ear. The IID is created when the intensity level of the stimulus in the better ear is decreased while maintaining a constant intensity level in the poorer ear. Training will begin at 50 dB above the SRT in the poorer ear (based on the DDT scores) and at 5 dB above the crossover point for the better ear (based on the DDT scores).

A total of five trials will be presented in a sequence and there will be 10 sequences per training session. Each of the 25 CVC words or digits 1 through 10 (excluding 7) will be presented to each ear during the session. The pairs will be randomized every time, and a word will never be paired with itself. After a sequence is completed, the difficulty of the task will be adjusted, in real time, based on performance on the prior task. If the child scored 4 or 5 of 5 correct in the poorer ear, then the IID will be decreased by 2 dB making the task more difficult. If the child scores 0, 1, or 2 of 5 correct, then the IID will be increased by 2 dB making the task easier. Last, if the child scores 3 of 5 correct, then the IID will remain unchanged for the next sequence.

One month following completion of DIID training, the child will be scheduled for both DDT and speech recognition in noise testing at the Division of Speech-Language and Hearing Therapy at Tygerberg Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants with delivery at >36 weeks gestation age
* Birth weight >2500g
* No major chromosomal anomalies, neural tube defects, seizures, HIV infection or other medical conditions that influenced neurodevelopmental outcomes and/or confounded the effects of ART and HIV exposure.

Exclusion Criteria:

* Child being older than the proposed age range
* Caregiver's or the child's refusal to participate

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Post Treatment Dichotic Digits Performance | Intervention will be 1-2 months
  A total of five trials will be presented in a sequence and there will be 10 sequences per training session. Each of the 25 consonant-vowel-consonant words or digits 1 through 10 (excluding 7) will be presented to each ear during the session. The pairs will be randomized every time, and a word will never be paired with itself. After a sequence is completed, the difficulty of the task will be adjusted, in real time, based on performance on the prior task. If the child scored 4 or 5 of 5 correct in the poorer ear, then the interaural intensity difference (IID) will be decreased by 2 dB making the task more difficult. If the child scores 0, 1, or 2 of 5 correct, then the IID will be increased by 2 dB making the task easier. Last, if the child scores 3 of 5 correct, then the IID will remain unchanged for the next sequence. Post treatment percent correct will be calculated and then compared to pre treatment percent correct.

IPD SHARING:
Plan to Share IPD: No